CLINICAL TRIAL: NCT02384603
Title: Effects of Two Physiotherapeutic Treatments in Pain and Posture of Fibromyalgia Patients: Randomized Controlled Trial
Brief Title: Effects of Physical Therapy in Pain and Posture of Fibromyalgia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Luciana Akemi Matsutani, PhD student, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 053/14
Record Dates: First submitted 2015-02-18; First posted 2015-03-10 (Estimated); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GPR and CBT (Experimental): Global postural reeducation associated with cognitive behavioral therapy; 01 session per week for 10 weeks
  Interventions: Other: Global postural reeducation; Other: Cognitive behavioral therapy
- SMSE and CBT (Active Comparator): Segmental muscle stretching exercises associated with cognitive behavioral therapy; 01 session per week for 10 weeks
  Interventions: Other: Segmental muscle stretching exercises; Other: Cognitive behavioral therapy

INTERVENTIONS:
Other: Global postural reeducation
  Arms: GPR and CBT
Other: Segmental muscle stretching exercises
  Arms: SMSE and CBT
Other: Cognitive behavioral therapy

SUMMARY:
The aim of this study is to compare the effects of two physiotherapeutic treatments of fibromyalgia: global postural reeducation associated with cognitive behavioral therapy and segmental muscle stretching exercises associated with cognitive behavioral therapy.

DETAILED DESCRIPTION:
Fibromyalgia is characterized mainly by chronic widespread pain. Segmental muscle stretching therapeutic exercises reduce the shortening of myofascial structures and recover the body flexibility. It is indicated for the treatment of chronic pain caused by osteo-myo-articular dysfunction. The pain behavior may be defined as the adoption of body postures and attitudes that a person communicates his/her pain. In this way, the global postural reeducation - a method of muscles chains stretching exercises - could be an important intervention. In addition, negative thoughts and dysfunctional beliefs are usual in situations of chronic pain, compromising the health recovery process. As part of a pain catastrophizing-related therapeutic approach, physiotherapist may help patients with chronic pain to develop positive, realistic and hope attitudes as based on the cognitive behavioral therapy model.

ELIGIBILITY:
Inclusion Criteria:

* Patients with fibromyalgia according to the 2010 American College of Rheumatology diagnostic criteria and the presence of at least 11 of 18 tender points.

Exclusion Criteria:

* Presence of joint deformities
* Independent walking disability
* Making another physiotherapeutic treatment at the same time.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-02; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Visual analogic scale of pain | 11 weeks

SECONDARY OUTCOMES:
McGill Pain Questionnaire | 11 weeks
Dolorimetry of the 18 tender points | 11 weeks
Survey of Pain Attitudes - brief version | 11 weeks
Body posture evaluation | 11 weeks
Modified Clinical Test of Sensory Interaction for Balance (CTSIBm) | 11 weeks
Sit-and-Reach Test | 11 weeks
Fibromyalgia Impact Questionnaire | 11 weeks
Narrative interview about self-care | 11 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Luciana A Matsutani, MSc, Principal Investigator — University of Sao Paulo; Amelia P Marques, PhD, Study Chair — University of Sao Paulo
Locations (1):
- Department of Physical Therapy, Speech and Occupational Therapy, School of Medicine of the University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Schmidt-Wilcke T, Clauw DJ. Fibromyalgia: from pathophysiology to therapy. Nat Rev Rheumatol. 2011 Jul 19;7(9):518-27. doi: 10.1038/nrrheum.2011.98. PMID 21769128
- [Background] Matsutani LA, Marques AP, Ferreira EA, Assumpcao A, Lage LV, Casarotto RA, Pereira CA. Effectiveness of muscle stretching exercises with and without laser therapy at tender points for patients with fibromyalgia. Clin Exp Rheumatol. 2007 May-Jun;25(3):410-5. PMID 17631737
- [Background] Teodori RM, Negri JR, Cruz MC, Marques AP. Global Postural Re-education: a literature review. Rev Bras Fisioter. 2011 May-Jun;15(3):185-9. English, Portuguese. PMID 21829981
- [Background] Campbell CM, McCauley L, Bounds SC, Mathur VA, Conn L, Simango M, Edwards RR, Fontaine KR. Changes in pain catastrophizing predict later changes in fibromyalgia clinical and experimental pain report: cross-lagged panel analyses of dispositional and situational catastrophizing. Arthritis Res Ther. 2012 Oct 25;14(5):R231. doi: 10.1186/ar4073. PMID 23098173
- [Derived] Matsutani LA, Sousa do Espirito Santo A, Ciscato M, Yuan SLK, Marques AP. Global posture reeducation compared with segmental muscle stretching exercises in the treatment of fibromyalgia: a randomized controlled trial. Trials. 2023 Jun 7;24(1):384. doi: 10.1186/s13063-023-07422-w. PMID 37280637